CLINICAL TRIAL: NCT03860922
Title: Conventional Magnetic Resonance Imaging Versus Magnetic Resonance Arthrography in Evaluation of Ankle Impingement Syndromes and Intra Articular Pathologies.
Brief Title: Conventional MRI Versus MR Arthrography in Evaluation of Ankle Impingement Syndromes and Intra Articular Pathologies.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Kawsar Abdel Halim Mohamed, principal Investigator, Assiut University
Other Study IDs: MRAAIS
Record Dates: First submitted 2019-02-23; First posted 2019-03-04 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2021-07

CONDITIONS: Ankle Impingement Syndrome
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Magnetic Resonance Imaging — all patient will undergo Magnetic resonance imaging and magnetic imaging arthrography of the ankle joint.

SUMMARY:
Chronic ankle pain is a common clinical problem with a wide differential diagnosis. Soft-tissue and osseous impingement syndromes are now increasingly recognized as a significant cause of chronic ankle pain. Ankle impingement syndromes are defined as pathologic conditions resulting in chronic, painful restriction to movement at the tibiotalar articulation secondary to soft-tissue or osseous abnormalities. Ankle impingement is classified according to its anatomic relationship to the tibiotalar joint as anterolateral, anterior, anteromedial, posteromedial, or posterior impingement.

DETAILED DESCRIPTION:
The anterolateral impingement syndrome is caused by obstruction of the so-called anterolateral gutter (ALG) or recess secondary to an inversion injury resulting in disruption of the syndesmotic and/or lateral collateral ligaments and capsule.

In anterior impingement,Arthroscopic evaluations suggest direct microtrauma to the talus and tibia as the aetiology. The natural course of this microtraumas to form osseous spurs.

In anteromedial impingement,The mechanism is not well understood but is likely a rare complication of a supination (inversion) injury rather than a pronation (eversion) injury as initially hypothesized.During the acute injury, there is damage to the anterior tibiotalar ligament, which subsequently thickens. In addition toligament thickening, osteophytes, synovitis and fractures have been described as other possible causative factors.

In posteromedial impingement, the common precipitating injury for posteromedial ankle impingement is a plantar flexion, inversion and internal rotation trauma. This can lead to damage to the PTTL and associated synovitis.

The majority of the posterior impingement syndromes are related to the posterior talus.The secondary ossification centre of the posterolateral talus forms around 8-13 years of age and then subsequently fuses within 1 year of that. Occasionally (approximately 7%), there may be non-fusion with a resultant ostrigonum.

Conventional MR imaging can accurately detect and localize osteophytes and associated lesions. In addition, MR imaging provides an easy evaluation of any articular cartilage changes, ligamentous injury, and occult bony contusions.

Direct magnetic resonance (MR) arthrography extends the capabilities of conventional MR imaging and utilizes the natural advantages gained from joint effusion. Contrast solution distends the joint capsule, outlines intra articular structures,and leaks into abnormalities.It can detect cartilage damage, intra articular loose bodies and osteochondral talar lesions.

ELIGIBILITY:
Inclusion Criteria:

* patients in different age groups and both sex referred from orthopedic outpatient clinic with chronic ankle pain and suspected clinically to have impingement syndrome.

Exclusion Criteria:

1. Inflammatory arthritis of ankle joint, infection in ankle joint, neoplasm around ankle joint.
2. Patients with contraindications for MRI, e.g. an implanted magnetic device, pacemakers or claustrophobia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients in different age groups and both sex clinically presented with chronic ankle pain.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-09-10 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Ligamentous disruption and thickening. | base line
  to detect the ligamentous disruption and thickening by conventional MRI and direct MR arthrography of the ankle joint.
Capsular thickening and synovitis. | baseline
  to detect the capsular thickening and synovitis by conventional MRI and direct MR arthrography of the ankle joint.

SECONDARY OUTCOMES:
correlate the findings of conventional MRI and MR Arthrography of the ankle with clinical and operative findings. | baseline
  to correlate the ligamentous disruption and thickening, capsular thickening and synovitis with clinical and operative findings (arthroscopy or open surgery).

CONTACTS AND LOCATIONS:
Overall Officials: Kawsar Mohamed, Principal Investigator — Assiut University
Locations (1):
- Faculty of medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Steinbach LS, Palmer WE, Schweitzer ME. Special focus session. MR arthrography. Radiographics. 2002 Sep-Oct;22(5):1223-46. doi: 10.1148/radiographics.22.5.g02se301223. PMID 12235350
- [Result] Mosier-La Clair SM, Monroe MT, Manoli A. Medial impingement syndrome of the anterior tibiotalar fascicle of the deltoid ligament on the talus. Foot Ankle Int. 2000 May;21(5):385-91. doi: 10.1177/107110070002100505. PMID 10830656
- [Result] Robinson P, White LM, Salonen D, Ogilvie-Harris D. Anteromedial impingement of the ankle: using MR arthrography to assess the anteromedial recess. AJR Am J Roentgenol. 2002 Mar;178(3):601-4. doi: 10.2214/ajr.178.3.1780601. PMID 11856682
- [Result] Donovan A, Rosenberg ZS. Extraarticular lateral hindfoot impingement with posterior tibial tendon tear: MRI correlation. AJR Am J Roentgenol. 2009 Sep;193(3):672-8. doi: 10.2214/AJR.08.2215. PMID 19696280
- [Result] Murawski CD, Kennedy JG. Anteromedial impingement in the ankle joint: outcomes following arthroscopy. Am J Sports Med. 2010 Oct;38(10):2017-24. doi: 10.1177/0363546510369335. Epub 2010 May 17. PMID 20479141
- [Result] Giannini S, Buda R, Mosca M, Parma A, Di Caprio F. Posterior ankle impingement. Foot Ankle Int. 2013 Mar;34(3):459-65. doi: 10.1177/1071100713477609. PMID 23520307
- [Result] Hayashi D, Roemer FW, D'Hooghe P, Guermazi A. Posterior ankle impingement in athletes: Pathogenesis, imaging features and differential diagnoses. Eur J Radiol. 2015 Nov;84(11):2231-41. doi: 10.1016/j.ejrad.2015.07.017. Epub 2015 Jul 17. PMID 26239710
- [Result] Paterson RS, Brown JN. The posteromedial impingement lesion of the ankle. A series of six cases. Am J Sports Med. 2001 Sep-Oct;29(5):550-7. doi: 10.1177/03635465010290050501. PMID 11573911
- [Result] Haller J, Bernt R, Seeger T, Weissenback A, Tuchler H, Resnick D. MR-imaging of anterior tibiotalar impingement syndrome: agreement, sensitivity and specificity of MR-imaging and indirect MR-arthrography. Eur J Radiol. 2006 Jun;58(3):450-60. doi: 10.1016/j.ejrad.2006.03.008. Epub 2006 Apr 18. PMID 16621392
- [Result] Robinson P, White LM, Salonen DC, Daniels TR, Ogilvie-Harris D. Anterolateral ankle impingement: mr arthrographic assessment of the anterolateral recess. Radiology. 2001 Oct;221(1):186-90. doi: 10.1148/radiol.2211001666. PMID 11568338